CLINICAL TRIAL: NCT05390606
Title: Pilot Study: Effects of Flourish HEC Vaginal Care System and BioGenesis Fertility Lubricant on Conception
Brief Title: Effects of Flourish HEC and BioGenesis to Improve Conception
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Vaginal Biome Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FRT0322
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Infertility; Infertility Unexplained
MeSH Terms: conditions — Infertility | interventions — Metabolism

STUDY DESIGN:
Intervention Model Description: A longitudinal open label randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control arm (No Intervention): Women follow routine care only, including prescribed medications and recommended techniques and supplements for attempting to become pregnant at home for up to three months.
- Flourish HEC + BioGenesis arm (Experimental): In addition to routine care followed by women in control arm, women in this arm also use the Flourish HEC (Hydroxyethylcellulose) vaginal care system and BioGenesis fertility lubricant for up to three months.
  Interventions: Combination Product: Flourish HEC and BioGenesis

INTERVENTIONS:
Combination Product: Flourish HEC and BioGenesis — Flourish HEC is a 3-component system, including: 1) Balance feminine wash, used daily; 2) BioNourish vaginal moisturizer, used daily before bed except if having intercourse; 3) BiopHresh homeopathic vaginal suppository with probiotics, used once every 3 days before bed except if having intercourse. BioNourish is a class II medical device with FDA 510k clearance, on the market for 2 years. BioGenesis is also a class II medical device with FDA 510k clearance, and is designated as a fertility lubricant, safe for sperm and embryos.
  Arms: Flourish HEC + BioGenesis arm

SUMMARY:
This study intends to address whether improving the vaginal microbiome can help couples increase chances of conceiving.

DETAILED DESCRIPTION:
Disrupted vaginal microbiomes are associated with a number of poor reproductive outcomes, including infertility, miscarriage, premature rupture of membranes, preterm labor and delivery, delivery of a low birthweight baby, and maternal infections (chorioamnionitis, endometritis). A healthy vaginal microbiome is typically thought to be one that is dominated by one of several Lactobacillus species, such as L. crispatus, L. gasseri, or L. jensenii. Several studies have shown that non-lactobacilli-dominant biomes are associated with poor in vitro fertilization or intrauterine insemination outcomes. Fewer studies have examined fertility in the home setting, and none to date has asked whether improving the vaginal microbiome (VMB) could increase fertility. This study addresses both. By assessing the VMB before and after using a vaginal care system which supports a healthy VMB, we will be able to examine whether there are associations between VMB composition and infertility, and whether shifting the VMB toward a lactobacillus-dominant state is able to improve chances of conception.

In this study, women will either follow routine care (control) or routine care plus the vaginal care system and fertility lubricant (intervention) for 3 months or until becoming pregnant, whichever comes first. In addition to tracking conception rates during those 3 months, we will follow women for an additional year following completion of the 3-month timeframe. If any woman is pregnant at the one-year mark, her pregnancy will be followed until delivery (or early termination) to track delivery outcomes and adverse events.

ELIGIBILITY:
Inclusion Criteria:

Women part of a cisgender couple aged 18 to 40 who are attempting to become pregnant and are attending a fertility clinic.

Exclusion Criteria:

1. Pregnant
2. Lactating
3. Severe male factor, hormonal imbalance (oligoovulatory/anovulatory cycles, cycles longer than 35 days), genetic abnormalities (chromosomal abnormality, common genetic mutation between partners), or severe uterine or tubal factor
4. Any diagnosis that would require the participant to undergo in vitro fertilization to become pregnant
5. Known allergies to any component of BioNourish®, Balance, BiopHresh®, or BioGenesis™
6. Known active vaginal infection at enrollment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Conception at home | 3 months
  Percentage of women becoming pregnant at home within the 3 month study.
Change in vaginal microbiome | Baseline to end of active study period, which is either at 3 months or upon confirmation of pregnancy, whichever occurs first.
  Vaginal microbiome composition tested by next-generation sequencing
Change in vaginal pH | Baseline to end of active study period, which is either at 3 months or upon confirmation of pregnancy, whichever occurs first.
  Vaginal pH tested by vaginal fluid applied to pH test strip

SECONDARY OUTCOMES:
Conception within one year | 15 months
  Percentage of women becoming pregnant by any method within the 3 month study or within one year after ending the study.
Rate of live birth | 24 months or fewer
  Percentage of women giving live birth within one year after ending the study; or if pregnant at one year, following to the end of her pregnancy.
Gestational age at delivery | 24 months or fewer
  Average gestational age of babies born within one year after ending the study; or if mothers are pregnant at one year, following to the end of her pregnancy.
Birthweight at delivery | 24 months or fewer
  Average weight of babies born within one year after ending the study; or if mothers are pregnant at one year, following to the end of her pregnancy.
Rates of pregnancy complications | 24 months or fewer
  Percentage of women experiencing complications (including preeclampsia, miscarriage/fetal loss/stillbirth, preterm/premature rupture of membranes, chorioamnionitis or endometritis, gestational diabetes, and any other adverse outcome) within one year after ending the study; or if mothers are pregnant at one year, following to the end of her pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Eyvazzadeh, MD, MS, MBA, Principal Investigator — Dr. Aimee Eyvazzadeh, Inc.
Locations (1):
- Dr. Aimee Eyvazzadeh, San Ramon, California, United States

IPD SHARING:
Plan to Share IPD: No